CLINICAL TRIAL: NCT04933097
Title: Evaluation of a New Screening Method for Sarcopenia in Rheumatoid Arthritis
Acronym: SARCO-RA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PA21032*
Record Dates: First submitted 2021-06-11; First posted 2021-06-21 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sarcopenia (Experimental): Only one arm with the sarcopenia assessment.
  Interventions: Device: Microfet2®

INTERVENTIONS:
Device: Microfet2® — Conducting a day hospitalization including analyses:
  1. Quantitative muscular analysis by measuring the DEXA of the whole body, the reference method for measuring body compartments and allowing the diagnosis of sarcopenia (IMMA<7 in men and 5.5 in women)
  2. Qualitative muscular analysis:
     * isokinetic measurement of muscular strength carried out on 3 muscle groups using a manual measurement sensor such as Microfet2 ® : quadriceps, triceps brachii, biceps
     * measurement of grip strength using Jamar® equipment validated as recommended by the EWGSOP
     * a walking test to assess the functional impact of sarcopenia and its severity

SUMMARY:
Evaluation of a new screening method for sarcopenia in rheumatoid arthritis

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is the most common inflammatory rheumatic disease, affecting 0.4-0.8% of the population. This inflammatory rheumatism leads to progressive, bilateral and symmetrical joint destruction, predominantly in the hands, which is responsible for significant functional repercussions, a sedentary lifestyle and a reduction in physical capacities leading to the onset of comorbidities. Among these comorbidities, sarcopenia is an emerging concept.

Sarcopenia is defined as a decrease in the quality and quantity of a person's muscles. It can be primary, and therefore due to physiological ageing, or secondary to a chronic disease such as inflammatory rheumatism. The definition of sarcopenia has become consensual since the 2019 European Working group on Sarcopenia in Older People (EWGSOP) recommendations and is characterised by:

* A decrease in strength. It is assessed by the grip test with a threshold of 27 kg in men and 16 kg in women. When this manual grip measurement is not possible, the authors advise measurement on an isokinetic device.
* a decrease in overall muscle mass. This is assessed either by dual energy X-ray absorptiometry (DEXA whole body, the reference technique) and defined by a decrease in the appendicular muscle mass index (AMMI) < 7 kg/m² in men and < 5.5 kg/m² in women (AMMI corresponds to the lean mass of the 4 limbs in relation to the height for Europeans); or on the scanographic measurement of the surface of the psoas muscle at L3.
* a decrease in muscular performance. This last point makes it possible to evaluate the severity of this sarcopenia. Muscular performance is assessed by walking speed and/or tests combining balance and walking such as the short physical performance battery test (SPPB) or the timed up and go (TUG).

The diagnosis of sarcopenia is certain when there is a decrease in muscle mass; it is characterised as severe when there is a decrease in physical performance.

Two other concepts are associated:

* Presarcopenia when there is a decrease in strength or muscle mass alone,
* Sarcopenic obesity when there is, in addition to the decrease in IMMA, an increase in the percentage of fat mass to 40% in women and 27% in men However, these tests are expensive, radiating and difficult to access for the general population. For these reasons, a screening algorithm is proposed by measuring hand grip strength, which is correlated with the decrease in overall muscle mass and physical performance in the general population.

The consequences of sarcopenia are numerous. In patients with severe sarcopenia, the risk of falling is doubled, increasing the risk of hospitalisation and the length of hospital stays. Severe sarcopenia is also associated with an earlier risk of death.

The prevalence of primary sarcopenia is between 15 and 20% in patients over 70 years of age, 40% after 80 years of age. In rheumatoid arthritis, Italian, Chinese, Japanese and Moroccan cohorts report a prevalence of sarcopenia in RA ranging from 21 to 40.9% with a median age of 52.3 to 56.5 years in these studies. There is thus an overrepresentation of this condition with an early age of onset compared to primary forms. In addition, there is pre-sarcopenia in 20% of cases.

This pre-sarcopenia could correspond to a window of opportunity for the management of these patients, both in terms of diet and rehabilitation. Indeed, the new recommendations of the European League Against Rheumatism concerning physical activity in inflammatory rheumatism propose the combination of aerobic and resistance work in patients with inflammatory rheumatism. However, when management is delayed, rehabilitation is sometimes no longer possible.

The specific consequence of sarcopenia in rheumatoid arthritis is a significant functional impact, with an increase in the Health Assessment Questionnaire (HAQ) score. In addition, loss of muscle mass and function was highly correlated with a decrease in overall bone mass, leading to a higher risk of osteoporotic fracture in this population. However, the method of assessing this sarcopenia does not seem to be the most appropriate in this population. There is a risk of overestimating the loss of strength through joint deformities. Indeed, one study showed that hand grip strength was correlated with age in the general population as opposed to a population of patients followed for RA. If this is not possible, the authors suggest that isokinetic measurements of other muscle groups should be performed to identify patients who may benefit from quantitative dynamometric muscle measurement.

There are several methods of assessing isokinetic strength. As muscle testing is very operator dependent, these new standardised and reproducible measurement techniques are expanding rapidly. There are two main types of dynamometry, isokinetic machines such as CYBEX® and BIODEX® and hand dynamometers, with a good correlation between the two techniques.

Because of its low cost, portability and ease of use, this technique could justify wider use, particularly in consultation. In this context of potential bias with overestimation of grip strength, it would be useful to evaluate isokinetic measurement of other muscle groups to assess which patients require quantitative muscle mass measurement.

However, no study has yet validated such a measure in rheumatoid arthritis. The hypothesis of our work is that manual dynamometry on other muscle groups would be more reproducible and reliable than grip force dynamometry for the detection of sarcopenia.

Primary endpoint:

Calculation of the sensitivity and specificity of quadriceps/triceps/biceps muscle strength measurement by handheld isokinetic dynamometer in screening for sarcopenia versus gold standard (DEXA whole body).

DEXA whole body is the gold standard method of measuring body compartments and allows the diagnosis of sarcopenia (IMMA<7 in men and 5.5 in women).

Manual dynamometry allows isokinetic measurements of muscle strength on 3 muscle groups using a manual measurement sensor of the Microfet2 ® type: quadriceps, triceps brachii, biceps (results in newtons/m²).

Both examinations will be performed during the patient's visit to the day hospital and will be interpreted blind to the results of each of these examinations.

Secondary endpoints:

1. Calculation of the intra-class correlation coefficient to assess inter-operator agreement for manual dynamometry. To evaluate the concordance, isokinetic measurements of muscle force on the 3 muscle groups using a manual measurement sensor such as Microfet2 ® will be performed by 2 different operators.
2. Comparison of the sensitivity and specificity values of the JAMAR® and Microfet2® dynamometer The isokinetic measurements of muscular force will be carried out using a Microfet2 ® type manual measurement sensor at the level of the quadriceps, triceps brachii, and biceps (results in newtons/m²) The measurement of grip strength will be performed with Jamar® equipment as recommended by the EWGSOP.

   DEXA whole body is the reference method for measuring body compartments and allows the diagnosis of sarcopenia (IMMA<7 in men and 5.5 in women).
3. Identification of risk factors for sarcopenia (smoking, alcohol, corticosteroids, duration of RA)
4. Description of comorbidities associated with sarcopenia (metabolic syndrome, cancer)
5. Impact on fatigue assessed by FSS questionnaire, HAQ assessment and SF 36

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis defined according to ACR/EULAR 2010 criteria,
* Follow-up at the University Hospital of Reims,
* Signed consent

Exclusion Criteria:

* Inability to perform a functional test (walking test)
* Patient under legal protection
* Patients not affiliated to the social security system
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Quadricepsmeasurement | Day 0
  The three measurements will be performed by two different operators and the results will be expressed in Newton/m.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided